CLINICAL TRIAL: NCT06518083
Title: The Relation Between Dynamic Change in Triglyceride- Glucose Index, Procalcitonin and Cardiac Affection in Patients Admitted to the Intensive Care Unit With Septic Shock.
Brief Title: The Relation Between Triglyceride- Glucose Index, Procalcitonin and Cardiac Affection in Septic Shock.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzi Ibrahim Mansour, Assistant -lecturer of critical care, Assiut University
Other Study IDs: 04-2024-100269
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group of patients with septic shock admitted to the ICU: The patients with septic shock admitted to the ICU will be observed for occurrence of cardiac events and their relation to triglyceride-glucose index and procalcitonin

SUMMARY:
The study is carried out to demonstrate the relation between Triglyceride -glucose index and cardiac affection in the patients admitted to the ICU with septic shock.

DETAILED DESCRIPTION:
Sepsis, a condition characterized by a dysregulated immune response to infection, is a prominent contributor to global mortality(1).

Insulin resistance (IR) is typified by reduced insulin sensitivity in peripheral tissues and is linked to various pathological conditions ( 2) The triglyceride-glucose (TyG) index, recognized as a surrogate marker of insulin resistance, has recently gained attention as a potential prognostic tool for various metabolic and cardiovascular diseases . ( 3) Preliminary investigations have revealed a correlation between metabolic disorders characterized by dysregulated lipid and glucose metabolism and the severity of sepsis. Notably, a high TyG index has been associated with increased in-hospital mortality in sepsis patients (4) studies only focused on the initial TyG value within the first 24 h of ICU admission and did not consider the dynamic changes in this marker over time. As insulin sensitivity in critically ill patients can change over time, (5) ,(6) It is possible that the TyG variability ratio (TyGVR) during hospital stay may be a better marker for adverse long-term prognosis and could be used for early risk stratification in critically ill patients, Procalcitonin (PCT) is produced during bacterial infections, sepsis, cardiogenic shock, major surgery, burns, multiple trauma, and after cardiac surgery( 7.8)

In this study we will discuss the relation between dynamic changes in both TyG index, procalcitonin and cardiac affection in the ICU patients admitted with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* 1- Adult patients (≥18 years) 2-Patients admitted to the ICU with septic shock.

Exclusion Criteria:

* 1-Patients who have mixed aetiology of shock. 2-Known previous cardiac disease ( cardiovascular disease, heart failure, arrhythmia )

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sample size calculation was carried out using G*Power 3 software (Faul et al., 2007) 1. A calculated minimum sample of 88 patients admitted to the ICU with septic shock will be needed to detect an effect size of 0.5 in the effect of TGD index variability on the cardiac affection in septic shock cases (OR 1.597; 95% CI 1.18 - 2.15)2, with an error probability of 0.05 and 80% power on a one-tailed test with normal x-distribution. The sample will be raised by 10% to compensate for dropouts, attrition and non-response to be 100 participants.
  1. Faul, F., Erdfelder, E., Lang, A.-G. & Buchner, A. (2007). G*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behavior Research Methods, 39, 175-191.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
1- To evaluate the effect of TyG index of on mortality of patients with septic shock.. | 3 months
  follow up the effect of elevated TyG index on increased mortality